CLINICAL TRIAL: NCT03508453
Title: A Phase 2, Randomised, Double-Blind, Placebo-Controlled Study of IC14 for Treatment of Patients With Rapidly Progressive Motor Neuron Disease
Brief Title: IC14 for Treatment of Amyotrophic Lateral Sclerosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study will not be conducted due to lack of funding
Sponsor: Implicit Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALS03
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2021-02

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease
Keywords: monoclonal antibody
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacy preparation of identical-appearing placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IC14 (monoclonal anti-CD14 antibody) (Active Comparator): IC14 4 mg/kg intravenously twice weekly for 12 weeks
  Interventions: Biological: IC14
- Placebo (Placebo Comparator): Placebo intravenously twice weekly for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: IC14 — Monoclonal antibody against CD14
  Arms: IC14 (monoclonal anti-CD14 antibody)
Other: Placebo — sterile normal saline for injection prepared to be identical to study drug
  Arms: Placebo

SUMMARY:
Fifty patients with amyotrophic lateral sclerosis that is progressing rapidly will be randomized to receive either the monoclonal antibody IC14 or placebo to be given intravenously over two hours twice weekly for 12 weeks. Blood and urine tests will be done to measure biomarkers in order to evaluate clinical response and to monitor for safety. Other evaluations include patient questionnaires about function, quality of life and mental function; pulmonary function test; and sniff nasal pressure.

DETAILED DESCRIPTION:
This will be a placebo-controlled, double-blind, parallel-group comparison.

Fifty patients with rapidly progressive ALS will be randomised to receive one of the following regimens:

* IC14 4 mg/kg given intravenously twice weekly for 12 weeks; or
* Identical-appearing placebo given intravenously twice weekly for 12 weeks. There will be an interim safety review by an independent Data Safety Monitoring Board after the initial 20 subjects have completed 4 weeks and 8 weeks of treatment. Study observation will continue until 12 weeks after the last dose of study drug.

The primary endpoint is:

• Treatment-related change in disease biomarker profiles [e.g., neurofilaments (Nf), urinary p75 neurotrophin receptor (p75NTR), cytokines, and soluble CD14].

The secondary endpoints are:

* Safety, tolerability and lack of immunogenicity of IC14.
* Treatment-related change in the Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R).
* Treatment-related change in respiratory function by seated forced vital capacity (FVC) parameters.
* Treatment-related change in inspiratory muscle strength by sniff nasal pressure (SNP) test.
* Treatment-related change in quality of life by the ALS Specific Quality of Life-Revised (ALSSQOL-R) score.
* Treatment-related change in cognitive function by Edinburgh Cognitive and Behavioural Assessment (ECAS) score.
* Treatment-related changes stratified by disease severity and prognostic indicators.
* Peak serum IC14 concentration following administration of the initial dose and peak serum concentration following a course of treatment.
* Area under the serum IC14 concentration versus time curve (AUC) following administration of the initial dose and following a course of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to initiation of any study-specific procedures.
2. Familial or sporadic MND defined as clinically possible, probable, or definite by Awaji-Shima Consensus Recommendations.
3. Rapidly progressive MND as defined by a decline of 3 or more points in the ALSFRS-R score during the prior 3 months.
4. First symptoms of MND within 3 years of informed consent.
5. Age between 18 and 75 years at time of informed consent.
6. Seated Forced Vital Capacity (FVC) ≥ 65% of predicted value.
7. Not taking riluzole or edaravone or on a stable dose of riluzole or edaravone for at least 3 months prior to screening visit.
8. Adequate bone marrow reserve, renal and liver function:

   * absolute neutrophil count ≥ 1.5 x 109/L
   * lymphocyte count < 6.0 x 109/L
   * platelet count ≥ 150 x 109/L
   * hemoglobin ≥ 110 g/L
   * eGFR ≥ 40 mL/min/1.73 m2
   * ALT and/or AST ≤ 2x ULN
   * total bilirubin ≤ 1.5x ULN
   * serum albumin ≥ 28 g/L
9. Females of childbearing potential should be using and committed to continue using one of the following acceptable birth control methods:

   * Sexual abstinence (inactivity) for 1 month prior to screening through study completion; or
   * Intrauterine device (IUD) in place for at least 3 months prior to study through study completion; or
   * Stable hormonal contraception for at least 3 months prior to study through study completion; or
   * Surgical sterilization (vasectomy) of male partner at least 6 months prior to study.
10. To be considered of non-childbearing potential, females should be surgically sterilized (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 2 months prior to study) or be post-menopausal and at least 3 years since last menses.
11. Males with female partners of childbearing potential must use contraception through study completion.
12. Able to give informed consent and able to comply with all study visits and all study procedures.

Exclusion Criteria:

1. Dependence on mechanical ventilation, defined as being unable to lay supine without it, unable to sleep without it, or continuous daytime use; presence of tracheostomy at screening; or presence of diaphragm pacing system at screening.
2. Treatment with a drug or device within the last 30 days that has not received regulatory approval.
3. Treatment within 12 months with immunomodulator or immunosuppressant agent (including but not limited to cyclophosphamide, cyclosporine, interferon-α, interferon-β-1a, rituximab, alemtuzumab, azathioprine, etanercept, infliximab, adalimumab, certolizumab, golimumab, anakinra, rilonacept, secukinumab, tocilizumab, mycophenolate mofetil, methotrexate, haematopoietic stem cell transplantation, anti-sense drugs, gene therapy, cell-depleting agents, total lymphoid irradiation). Treatment with intravenous immunoglobulin within 2 months or dimethyl fumarate within 3 months. Non-steroidal anti-inflammatory drugs are acceptable.
4. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other opportunistic infections; or major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks.
5. Live-attenuated vaccines within 30 days before dosing. Subjects must agree to forego live-attenuated vaccines throughout the study, including 12 weeks after the last dose of study drug.
6. History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies.
7. Presence of any of the following clinical conditions:

   * History of one or more of the following: cardiac insufficiency (New York Heart Association [NYHA] III/IV), uncontrolled cardiac arrhythmias, unstable ischemic heart disease, or uncontrolled hypertension (systolic blood pressure > 170 mmHg or diastolic blood pressure > 110 mmHg).
   * History of venous thromboembolic disease within 12 months, myocardial infarction, or cerebrovascular accident.
   * Unstable pulmonary, renal, hepatic, endocrine or hematologic disease.
   * Autoimmune disease, mixed connective tissue disease, scleroderma, polymyositis, or significant systemic involvement secondary to rheumatoid arthritis.
   * Evidence of active malignant disease, malignancies diagnosed within the previous 5 years, or breast cancer diagnosed within the previous 5 years (except skin cancers other than melanoma).
   * History of human immunodeficiency virus infection or other immunodeficiency illness.
   * Unstable psychiatric illness defined as psychosis or untreated major depression within 90 days.
   * History of drug abuse (not including marijuana use) or alcoholism within the past 12 months.
   * Significant neuromuscular disease other than MND.
   * Other ongoing disease that may cause neuropathy, such as toxin exposure, dietary deficiency, uncontrolled diabetes, hyperthyroidism, cancer, systemic lupus erythematosus or other connective diseases, infection with HIV, hepatitis B virus (HBV), or hepatitis C (HCV), Lyme disease, multiple myeloma, Waldenström's macroglobulinemia, amyloid, and hereditary neuropathy.
8. Pregnancy or breastfeeding.
9. Deprivation of freedom by administrative or court order.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-15 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Neurofilament (biomarker) | 12 weeks
  Treatment-related change in concentration of neurofilament (picograms per milliliter)
Urinary p75 neurotrophin receptor (biomarker) | 12 weeks
  Treatment-related change in concentration of urinary p75 neurotrophin receptor (nanograms per milligram creatinine)
Monocyte CD14 receptor occupancy | 12 weeks
  Treatment-related change in percent monocyte receptor occupancy

SECONDARY OUTCOMES:
Functional status | 12 weeks
  Treatment-related change in Revised Amyotrophic Lateral Sclerosis Functional Rating Scale [0 (worst) to 48 (best)]
Respiratory function | 12 weeks
  Treatment-related change in percent normal Forced Vital Capacity [0% (worst) to 100%(best)]
Muscle function | 12 weeks
  Treatment-related change in percent normal Sniff Nasal Pressure [0% (worst) to 100% (best)]
Quality of life measured by ALSSQOL | 12 weeks
  Treatment-related change in Amyotrophic Lateral Sclerosis Specific Quality of Life - Revised questionnaire [0 (worst) to 460 (best)]
Cognitive and behavioural assessment | 12 weeks
  Treatment-related change in Edinburgh Cognitive and Behavioural Assessment Score [0(worst) to 136 (best)]
Maximum plasma concentration (Cmax) | 12 weeks
  Maximum serum IC14 concentration (micrograms per milliliter)
Area under the curve | 12 weeks
  Area under the curve for serum IC14 (microgram x hr/mL)
Immunogenicity | 16 weeks
  Development of human anti-monoclonal antibodies following treatment
Adverse events (safety, tolerability) | 16 weeks
  Incidence of treatment-emergent adverse events (safety, tolerability) classified by MedDRA

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Henderson, MBBS, Study Chair — Royal Brisbane & Women's Hospital
Locations (1):
- Royal Brisbane and Women's Hospital, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No